CLINICAL TRIAL: NCT02301741
Title: Using an Interactive Game to Reduce Fear & Increase Spine Motion in Low Back Pain
Brief Title: Using an Interactive Game to Reduce Fear and Increase Spine Motion in Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: R21AR064430-01A1 (NIH)
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Low Back Pain
Keywords: chronic low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Game Condition (Experimental): Participants in the GAME condition will complete laboratory sessions on five consecutive days. Session 1 (baseline) and Session 5 (post-test) will be used to assess lumbar spine motion and expectations of pain and harm during standardized reaching tasks. In sessions 2 through 4 they will play the virtual dodge ball game.
  Interventions: Behavioral: Game
- Control Condition (No Intervention): Participants in the CONTROL condition will complete baseline and post-test standardized reaching tasks, but will not play the game in the intervening three days.

INTERVENTIONS:
Behavioral: Game — We will assess the influence of participation in a computer game of virtual dodge ball that requires whole-body reaching movements to manipulate an on-screen avatar. We will gradually reduce the gain of lumbar spine motion of the participant's on-screen avatar across the three game sessions such that participants will need to produce progressively larger excursions of the lumbar spine to manipulate their avatar's spinal motion. Specifically, in game session 1, the spine motion of the avatar is equal to that of the participant (gain=1); in session 2 spine motion of the avatar is 5% less than the participant (gain=0.95); in session 3 spine motion of the avatar is 10% less than the participant (gain=0.90).
  Arms: Game Condition

SUMMARY:
A fundamental clinical problem in individuals with chronic low back pain is the significant alteration in movement patterns that restrict lumbar spine motion. This is particularly true for individuals with fear of re-injury with movement (i.e., kinesiophobia). The primary aims of the current study are to use a whole body video game environment to 1) determine the effects of game play on lumbar spine flexion and expectations of pain and harm and 2) determine the effects of altered movement gain on lumbar spine flexion.

DETAILED DESCRIPTION:
Using a 2 groups (Game, Control) between subjects design, the investigators will assess the influence of participation in a computer game of virtual dodge ball that requires whole-body reaching movements to manipulate an on-screen avatar. Further, the investigators will gradually reduce the gain of lumbar spine motion of the participant's on-screen avatar across the three game sessions such that participants will need to produce progressively larger excursions of the lumbar spine to manipulate their avatar's spinal motion. Specifically, in game session 1, the spine motion of the avatar is equal to that of the participant (gain=1); in session 2 spine motion of the avatar is 5% less than the participant (gain=0.95); in session 3 spine motion of the avatar is 10% less than the participant (gain=0.90). The investigators will recruit participants with chronic low back pain and kinesiophobia. Participants in the GAME condition will complete laboratory sessions on five consecutive days. Session 1 (baseline) and Session 5 (post-test) will be used to assess lumbar spine motion and expectations of pain and harm during standardized reaching tasks. In sessions 2 through 4 they will play the virtual dodge ball game. Participants in the CONTROL condition will complete baseline and post-test standardized reaching tasks, but will not play the game in the intervening three days.

ELIGIBILITY:
Inclusion Criteria:

1. Answer Yes to the following:

   * Have you had low back pain constantly or on most days for the last 3 months?
   * Has your back pain caused you to seek medical care?
2. Low back pain is classified from category 1 (back pain that does not radiate) through category 3 (back pain that radiates beyond the knee, but without neurological signs) on the Classification System of the Quebec Task Force on Spinal Disorders.
3. Report elevated levels of kinesiophobia.
4. Report no health conditions that may restrict movement or preclude safe participation.

Exclusion Criteria:

Individuals must not:

1. Have a personal history of the following neurological disorders: Alzheimer's, Amyotrophic Lateral Sclerosis, Multiple Sclerosis, Parkinson's, Stroke
2. Have a personal history of the following cardiorespiratory disorders: Congestive heart failure, Heart attack in past 24 months
3. Have a personal history of the following musculoskeletal disorders: Rheumatoid Arthritis, pathologic fractures of the spine, avascular necrosis or osteonecrosis, severe osteoarthritis.
4. Have a personal history of spine surgery or a hip arthroplasty
5. Have active cancer or recent, unexplained weight loss
6. Report being blind
7. Report being pregnant
8. Report current or pending litigation related to back pain
9. Currently be taking narcotic medication
10. Score in the clinically significant range for substance abuse (Drug Abuse Screening Test (DAST) > 6), alcohol abuse (Alcohol Use Disorders Identification Test (AUDIT-C) > 4), or depression (Center for Epidemiological Studies-Depression (CES-D) > 16).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Lumbar spine flexion changes | baseline (day 1) to post-test (day 5)
  This assessment tracks the magnitude of spine motion used to complete standardized reaching tasks in which participants reach to 3 targets (High, Middle, Low) located in the mid-sagittal plane. Participants will perform five reaching trials to each the target location and then return to an upright posture, with rest provided between each trial. Lumbar spine flexion will be defined as the change in joint angle (i.e., the difference between the joint angles at the beginning of the trial before the go signal and those extracted 100 ms after target contact). The average of the five reaches to each target location will serve as the dependent variable.
Expectation of pain changes | baseline (day 1) to post-test (day 5)
  For each target height, prior to the first reaching trial participants will be asked to rate the level of "expected pain" using a visual analog scale. The scale will consist of a 10-cm horizontal line with no numbers, marks, or descriptive vocabulary along its length. The scale will be anchored with the descriptors "No pain" and "Worst pain imaginable", respectively, at each end of the line. The pain expectancy ratings for each target location will serve as the dependent variable.
Expectation of harm changes | baseline (day 1) to post-test (day 5)
  For each target height, prior to the first reaching trial participants will be asked to rate the level of "expected harm" using a visual analog scale. The scale will consist of a 10-cm horizontal line with no numbers, marks, or descriptive vocabulary along its length. The scale will be anchored with "Not at all concerned" and "Extremely concerned" regarding potential harm to the back during task performance. The harm expectancy ratings for each target location will serve as the dependent variable.

SECONDARY OUTCOMES:
Lumbar spine flexion change as a function of altered movement gain | session day 2, 3 and 4
  Change in lumbar flexion measured during game play will be measured across the three gaming sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

REFERENCES:
- [Derived] Thomas JS, France CR, Applegate ME, Leitkam ST, Walkowski S. Feasibility and Safety of a Virtual Reality Dodgeball Intervention for Chronic Low Back Pain: A Randomized Clinical Trial. J Pain. 2016 Dec;17(12):1302-1317. doi: 10.1016/j.jpain.2016.08.011. Epub 2016 Sep 9. PMID 27616607